CLINICAL TRIAL: NCT02810847
Title: The Use of Interactive Binocular Treatment (I-BiT) for the Management of Anisometropic, Strabismic and Mixed Amblyopia in Children Aged 3.5 - 12 Years
Acronym: I-BiT Plus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13OY006
Record Dates: First submitted 2016-04-26; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Amblyopia; Strabismus
Keywords: Amblyopia; strabismus; virtual reality; computer games
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-BiT Plus (Experimental): 6 weeks of I-Bit treatment plus (at least 30 mins/day, 6 days/week)
  Interventions: Device: I-Bit plus
- Control (No Intervention): Refractive adaption or observation

INTERVENTIONS:
Device: I-Bit plus — The study will treat amblyopia (lazy eye) using 3-D computer technology and active shutter glasses. Computer games and DVD's are viewed through the active shutter glasses and are specially prepared to preferentially stimulate the lazy eye; the child can only play the game accurately if they are using their lazy eye.
  Arms: I-BiT Plus

SUMMARY:
Around one child in fifty has a lazy eye (termed amblyopia) where the eye is structurally normal but the vision fails to develop correctly. Around half of these children also have a squint (strabismus) where each eye has a different direction of gaze. This condition is the commonest cause of visual impairment in one eye in children.

This is a randomised control trial of wearing glasses alone (which will result in some visual improvement, termed refractive adaptation) and wearing glasses combined with using I-BiT Plus.

The hypothesis is that using I-BiT Plus will result in an improved visual outcome.

DETAILED DESCRIPTION:
This study will treat amblyopia (lazy eye) using 3-D computer technology and active shutter glasses. Computer games and DVD's are viewed through the active shutter glasses and are specially prepared to preferentially stimulate the lazy eye; the child can only play the games accurately if they are using their lazy eye. The study is funded by the NIHR and will be undertaken as a randomised control trial to compare this against normal computer games and DVD viewing combined with continuing refractive adaptation (a process that is known to occur for up to 30 weeks). Patients will receive 6 weeks of treatment (recommended 30 mins minimum of play time per day for 6 weeks in the treatment arm) and level of vision will be assessed after 6 weeks and the visual improvement (they will be wearing glasses and also undergoing refractive adaptation) compared with the control. Patients will return to standard care after the trial period which, at 6 weeks, should not affect the final visual outcome in a negative way. The participants will be recruited from patients currently attending one of the 4 trial sites and will have a diagnosis of amblyopia, and be aged between 3 years 6 months and 9 years 11 months. Current treatments for amblyopia include wearing an eye patch over the good eye for up to 6 hours per day, or using eye drops to blur the image in the good eye for periods of 4 weeks at a time. The aim is both to avoid the need for patching or penalisation (which are unpopular treatments) and to get an improved visual outcome.

Assessment study: A study on 62 patients where the investigators will compare the visual acuity, angle of strabismus, stereoacuity and depth of suppression as estimated by I-BiT against measurements made at orthoptic assessment. This data will help interpret the results of the randomised controlled trial and help direct future development.

ELIGIBILITY:
Inclusion Criteria:

* The child must be aged between 3 years 6 months and 9 years 11 months (upper limit is one day before their 10th birthday on day of consent.)
* Visual acuity difference of at least 0.3 log units, with the amblyopic eye being 0.3 logMAR or worse.
* Must have undergone a minimum of 12 weeks refractive adaptation.
* Those in group one must not have had patching or penalisation at all previously but the other two groups' participants may have had previous occlusion.
* Must not have had previous strabismus surgery (for groups one and two, and for group three, they must start the treatment within 4 weeks of having surgery.
* Must be able to use the I-BiT plus system.

Exclusion Criteria:

* Stimulus deprivation amblyopia.
* Other ocular or neurological disease affecting the visual system (including Down's syndrome, developmental delay,Craniofacial syndrome,Foetal Alcohol Syndrome, and cerebral palsy among other conditions).
* Photosensitive epilepsy.
* Parent, guardian or child not prepared to give consent.

Ages: 42 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of visual acuity from baseline to week six post randomisation visit between the two arms in each group. | 6 weeks

SECONDARY OUTCOMES:
Successful delivery and installation of equipment to patients' homes, and any reasons for failure | 10 weeks
The ability of the patients to use the equipment in their home (unsupervised) setting and any reasons why not. Ocular alignment Stereoacuity Proportion of patients completing course | 10 weeks
The time taken by the patients to use the equipment in their home (unsupervised) setting. | 10 weeks
The robustness of the equipment by measuring failure / breakage rate. | 10 weeks
Completeness of outcome measures will be assessed via the frequency of missing data. | 10 weeks
The recruitment rate and reasons for not taking part. | 10 weeks
The retention rate and reasons for drop out. | 10 weeks
Any problems encountered with the randomisation process. | 10 weeks
The standard deviation in visual acuity at 6 weeks; this will inform sample size calculations for a future trial to assess effectiveness of the I-BiT™ system. | 6 weeks
Change in visual acuity in the amblyopic eye from baseline to weeks 3 and 10 post randomisation between the two arms. | 8 Weeks
Change in stereoacuity from baseline to week 3 post randomisation between the two arms. | 3 weeks
Change in stereoacuity from week 3 to weeks 6 and 10 for the I-BiT treated groups. | 8 Weeks
Change in binocular status and ocular alignment from baseline to week 6 post randomisation between the two arms in each group. | 6 Weeks
Change in binocular status and ocular alignment from week 6 to week 10 for the I-BiT treated groups. | 5 weeks
Quality of life questionnaire at week 6. | 6 weeks
Proportion of patients completing course of treatment (defined as minimum of 18 hours in total, which equates to 30 minutes per day 6 days per week for six weeks). | 18 hours
The change in visual acuity, and angle of strabismus between weeks 3, 6 and 10 for the I-BiT treated groups. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander JE Foss, DM FRCOphth MRCP, Principal Investigator — Nottingham University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown R, Blanchfield P, Fakis A, McGraw P, Foss AJE; I-BiT Study Group. Clinical investigation plan for the use of interactive binocular treatment (I-BiT) for the management of anisometropic, strabismic and mixed amblyopia in children aged 3.5-12 years: a randomised controlled trial. Trials. 2019 Jul 16;20(1):437. doi: 10.1186/s13063-019-3523-0. PMID 31311577